CLINICAL TRIAL: NCT07229365
Title: Children's Viewing Behavior in Myopia Control Spectacles
Brief Title: Children's Viewing Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPRO-2507-002
Record Dates: First submitted 2025-11-12; First posted 2025-11-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Myopia Progression; Juvenile Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SightGlass Vision Test Arm 1 (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Novel spectacle lens design
- SightGlass Vision Test Arm 2 (Experimental): Single vision, impact-resistant spectacle lenses
  Interventions: Device: Spectacle lenses

INTERVENTIONS:
Device: Novel spectacle lens design — Use of lenses may reduce the rate of progression of juvenile myopia
  Arms: SightGlass Vision Test Arm 1
Device: Spectacle lenses — Use of lenses may reduce the rate of progression of juvenile myopia
  Arms: SightGlass Vision Test Arm 2

SUMMARY:
The aim of this study is to investigate the area of the spectacle lens in which a subject is viewing through regardless of task being performed.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is 7-14 years of age, inclusive
* Requires spherical spectacle lenses within the power range available for the study lenses
* Parent/guardian has read and understood the informed consent form, and the child has provided age-appropriate assent
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best corrected
* Has had a self-reported oculo-visual examination in the last two years
* Spectacle cylinder of ≤ -0.75DC in both eyes

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Is unable to complete the necessary study activities
* Has any systemic disease affecting ocular health
* Is using any systemic or topical medications (including pharmaceutical myopia control therapy) that will affect ocular health
* Is aphakic

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Activity dependent, gaze location in myopia control spectacles | 2 months
Subjective/objective quantification of activity via survey or observation | 2 months
Pupil size | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States